CLINICAL TRIAL: NCT04983069
Title: Neonatal Outcome of Children With Antenatal Colic Hyperechogenicity
Acronym: COLONECHOGENE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0376
Record Dates: First submitted 2021-07-05; First posted 2021-07-30 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Colic; Nephropathy
Keywords: Gynecology-Obstetrics; Ultrasound; Medical genetics; Pediatrics; Nephropathy; Colic hyperechogenicity; Antenatal; Lysinuria-cystinuria; lysinuric protein intolerance
MeSH Terms: conditions — Colic; Kidney Diseases; Lysinuric Protein Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal colic hyper-echogenicity is a presenting symptoms for cystinuria lysinuria.

A few cases of fetuses with dibasic protein intolerance (more complex prognosis) presented with colic hyper-echogenicity antenatal.

The aim of this retrospective study is to assess the outcome of fetuses with colic hyperechogenicity in order to increase prenatal counseling

DETAILED DESCRIPTION:
Observational multicenter retrospective study from january 2011 to january 2021.

No supplementary visit, directly related to the research, will be necessary. This study does not change the usual management of the patient.

Patients will be included after their usual medical check-up.

ELIGIBILITY:
Inclusion criteria:

* Fetuses with prenatal colic hyperechogenicity
* Between January 2011 and January 2021
* Born without term limitation.

Exclusion criteria:

* Intestinal hyperechogenicity
* polymalformative syndrome
* Patients Age<15 years

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Foetuses with prenatal colic hyperechogenicity
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Postnatal outcome of fetuses | day 1 (End of follow up)
  Postnatal outcome of fetuses with hyperechogenic colon.

SECONDARY OUTCOMES:
Rate of lysinuria/cystinuria | day 1 (End of follow up)
  Rate of lysinuria/cystinuria
Rate of dibasic protein intolerance | day 1 (End of follow up)
  Rate of dibasic protein intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC